CLINICAL TRIAL: NCT05164588
Title: A Prospective Study of Traumatic Eye Injuries in the Period From January 2022 to June 2022 in Sohag University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Safaa Lotfy Ali, Teaching assistant in Forensic Medicine and Clinical Toxicology, Sohag University
Other Study IDs: Soh-Med-21-12-02
Record Dates: First submitted 2021-12-12; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Eye Injuries
MeSH Terms: conditions — Eye Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Statistics — Study and analyze the medicolegal aspects of different eye trauma cases ( patterns of injuries, mechanisms, causes, site of trauma and outcome)

SUMMARY:
Ocular trauma is one of the main causes of severe ocular morbidity. It represents a serious public health problem and leading cause of visual impairment. It is an important and preventable cause of visual impairment in both developing and developed countries.

ELIGIBILITY:
Inclusion Criteria:

* All diagnosed cases of eye trauma, regardless of gender, laterality, duration of presentation and other chronic systemic illness

Exclusion Criteria:

* patients with previous history of eye trauma or other pathological condition affecting visual acuity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All diagnosed cases of eye trauma, regardless of gender, laterality, duration of presentation and other chronic systemic illness
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate eye trauma cases at Sohag University Hospitals through statistical methods | 6 months
  We will analyze data about participants, mechanism of injuries, site of trauma and if the time of arrival if delayed or certain treatment will affect the outcome and then we will determine the causes of better outcome to improve the outcome of future cases

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mir TA, Canner JK, Zafar S, Srikumaran D, Friedman DS, Woreta FA. Characteristics of Open Globe Injuries in the United States From 2006 to 2014. JAMA Ophthalmol. 2020 Mar 1;138(3):268-275. doi: 10.1001/jamaophthalmol.2019.5823. PMID 31971539
- [Background] Matsa E, Shi J, Wheeler KK, McCarthy T, McGregor ML, Leonard JC. Trends in US Emergency Department Visits for Pediatric Acute Ocular Injury. JAMA Ophthalmol. 2018 Aug 1;136(8):895-903. doi: 10.1001/jamaophthalmol.2018.2062. PMID 29879287
- [Background] Low L, Hodson J, Morris D, Desai P, MacEwen C. Socioeconomic deprivation and serious ocular trauma in Scotland: a national prospective study. Br J Ophthalmol. 2017 Oct;101(10):1395-1398. doi: 10.1136/bjophthalmol-2016-309875. Epub 2017 Mar 8. PMID 28274942